CLINICAL TRIAL: NCT02941549
Title: A Randomised, Double-Blind, Placebo-Controlled, Exploratory Phase IIa Study To Assess The Safety And Efficacy Of Orally Administered Epeleuton In NAFLD Patients.
Brief Title: Safety And Efficacy Study Of Orally Administered Epeleuton In Patients With NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afimmune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DS102A-02; 2016-000311-33 (EudraCT Number)
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Results first posted 2022-04-21 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Non Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — epeleuton

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): 2 x placebo 500 mg capsules orally administered twice a day (4 capsules daily) for 16 weeks
  Interventions: Other: Placebo capsules
- 1000 mg Epeleuton (Experimental): 1 x Epeleuton 500 mg capsule and 1 x placebo 500 mg capsule orally administered twice a day (4 capsules daily) for 16 weeks
  Interventions: Drug: Epeleuton
- 2000 mg Epeleuton (Experimental): 2 x Epeleuton 500 mg capsules orally administered twice a day (4 capsules daily) for 16 weeks
  Interventions: Drug: Epeleuton

INTERVENTIONS:
Other: Placebo capsules
  Arms: Placebo
Drug: Epeleuton
  Arms: 1000 mg Epeleuton; 2000 mg Epeleuton

SUMMARY:
The purpose of this randomised, double-blind, placebo-controlled, parallel group study is to assess the safety and efficacy of orally administered Epeleuton capsules versus placebo in the treatment of adult patients with Non Alcoholic Fatty Liver Disease (NAFLD)

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with NAFLD by the presence of hepatic steatosis on imaging or histology in the absence of any secondary causes.
2. Patients with an ALT ≥ 1.5 upper limit of normal (ULN) and < 5 ULN on two occasions 7 or more days apart during screening.
3. Patients with historical liver biopsy showing NASH and/or ≥ F1 fibrosis OR NFS ≥ -1.455 OR Fib- 4 ≥ 1.3 OR Fibroscan ≥8kPa within 3 months of screening.
4. Patients with a body mass index (BMI) between 25.0 and 40.0 kg/m² inclusive. Patients with a history of controlled obesity or controlled diabetes are allowed on the study.
5. Patients whose pre-study clinical laboratory findings do not interfere with their participation in the study, in the opinion of the Investigator.
6. Patients aged between 18 and 75 years inclusive.
7. Female patients and male patients with female partners of child bearing potential must use adequate contraception or have a sterilized partner for the duration of the study. Adequate contraception is defined as: systemic hormonal contraceptives; intrauterine device or barrier method of contraception in conjunction with spermicide; or agree to sexual abstinence, defined as a patient refraining from heterosexual intercourse during the entire period of risk associated with the study treatments and in line with their preferred and usual lifestyle. Hormonal contraceptives must be on a stable dose for at least one month before baseline.
8. Patients who are able to communicate well with the Investigator, to understand and comply with the requirements of the study, and understand and sign the written informed consent.

Exclusion Criteria:

1. Patients with an unstable metabolic condition such as weight change > 5% in the 3 months prior to inclusion.
2. Patients with medical/surgical history of gastric bypass surgery, orthotopic liver transplant (OLT) or listed for OLT.
3. Patients with uncontrolled diabetes mellitus type 2, i.e. HbA1c ≥ 9% (75 mmol/mol) at the time of screening.
4. Patients with decompensated or severe liver disease as evidenced by one or more of the following: confirmed cirrhosis or suspicion of cirrhosis, esophageal varices, ascites, suspicion of portal hypertension, hospitalization for liver disease within 60 days of screening, bilirubin ≥ 2 x ULN, or ALT or AST ≥ 5 x ULN. Patients with Gilbert's syndrome are eligible if the conjugated bilirubin is ≤ 1.5 x ULN.
5. Patients with inflammatory bowel disease that is either active or requiring medical therapy.
6. Patients with diagnosed or suspected autoimmune diseases such as systemic lupus erythematosus and/or rheumatoid arthritis.
7. Patients with a history of or active non-liver malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas).
8. Patients with a significant systemic or major illness other than liver disease, including coronary artery disease, cerebrovascular disease, pulmonary disease, renal insufficiency, serious psychiatric disease, respiratory or hypertensive disease, as well as diabetes and arthritis that, in the opinion of the Investigator, would preclude the patient from participating in and completing the study.
9. Patients requiring anti-diabetic treatment (including insulin sensitizing agents), and/or lipid lowering treatment, and who are not on a stable dose for at least 3 months prior to screening should be excluded. If patients are insulin dependent this treatment should have commenced at least 3 months prior to screening, however changes in dose are permitted.
10. Patients with known hypersensitivity to any ingredients of the study treatment.
11. Patients with a positive test for human immunodeficiency virus antibodies, Hepatitis B surface antigen or Hepatitis C antibodies at screening.
12. Patients with liver disease of other etiologies such as drug-induced, autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, haemochromatosis, alpha-1 antitrypsin deficiency or Wilson's disease.
13. Patients with a significant history of drug/solvent abuse, in the opinion of the investigator.
14. Patients with a history of alcohol abuse in the opinion of the Investigator, or who currently drinks in excess of 21 units per week (males) or 14 units per week (females), whereby a unit consists of 10ml or 8mg of pure alcohol.
15. Patients who have used dietary supplements rich in omega-3 or omega-6 fatty acids in the 4 weeks prior to baseline.
16. Patients who have participated in any other clinical study with an investigational drug within 3 months before the first day of administration of study treatment.
17. Patients who are pregnant, planning pregnancy, breastfeeding and/or are unwilling to use adequate contraception (as specified in inclusion criterion 7) during the study.
18. Patients, in the opinion of the Investigator, not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Newsome, MBChB, FRCPE, Ph.D, Principal Investigator — University of Birmingham
Locations (16):
- Georgia (3):
  - Georgia Site 1, Kutaisi
  - Georgia Site 2, Kutaisi
  - Georgia Site 3, Tbilisi
- Ukraine (4):
  - Ukraine Site 3, Dnipro
  - Ukraine Site 1, Kharkiv
  - Ukraine Site 2, Kyiv
  - Ukraine Site 4, Kyiv
- United Kingdom (9):
  - UK Site 1, Birmingham, UK
  - UK Site 5, Birmingham, UK
  - UK Site 6, London, UK
  - UK Site 7, Norwich, UK
  - UK Site 3, Oxford, UK
  - UK Site 4, Plymouth, UK
  - UK Site 2, Portsmouth, UK
  - UK Site 9, Belfast
  - UK Site 8, Liverpool

REFERENCES:
- [Derived] Climax J, Newsome PN, Hamza M, Weissbach M, Coughlan D, Sattar N, McGuire DK, Bhatt DL. Effects of Epeleuton, a Novel Synthetic Second-Generation n-3 Fatty Acid, on Non-Alcoholic Fatty Liver Disease, Triglycerides, Glycemic Control, and Cardiometabolic and Inflammatory Markers. J Am Heart Assoc. 2020 Aug 18;9(16):e016334. doi: 10.1161/JAHA.119.016334. Epub 2020 Aug 11. PMID 32779505

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 96 patients were randomised in a 1:1:1 ratio.
Groups:
- 2000mg Epeleuton: 2 x Epeleuton 500 mg capsules orally administered twice a day (4 capsules daily) for 16 weeks
Period: Overall Study
Arm/Group | Placebo | 1000 mg Epeleuton | 2000mg Epeleuton
Started | 31 | 32 | 33
Completed | 28 | 31 | 31
Not Completed | 3 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all randomised patients who received at least one administration of study treatment and have at least one post-baseline measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton | Total
Number analyzed (Participants) | 31 | 32 | 33 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.67) | 50.8 (13.72) | 46.1 (11.92) | 48.4 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 12 | 33
  Male | 22 | 20 | 21 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 28 | 30 | 33 | 91
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum ALT (Alanine Aminotransferase) From Baseline to Week 16
Description: Change in serum ALT from baseline to Week 16 using ANCOVA.
Time Frame: 16 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 30 | 32 | 31
U/L | -16.3 [-44.2 to 11.7] | -6.9 [-34.5 to 20.7] | -10.1 [-36.9 to 16.8]
Statistical Analysis 1: Comparison: Placebo vs 1000 mg Epeleuton; Test type: Superiority; p = 0.5946, ANCOVA; LS Mean Difference = -6.9, 95% CI 2-sided [-34.5 to 20.7]
Statistical Analysis 2: Comparison: Placebo vs 2000 mg Epeleuton; Test type: Superiority; p = 0.7309, ANCOVA; LS Mean Difference = -10.1, 95% CI 2-sided [-36.9 to 16.8]

2. Primary Outcome: Change in Liver Stiffness Measurements by Transient Elastography From Baseline to Week 16
Description: To evaluate change in liver stiffness measurements using Transient Elastography from baseline to Week 16 using FibroScan® 502 Touch model or equivalent.
Time Frame: 16 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 30 | 32 | 31
kPa | -2.226 [-3.07 to -1.38] | -1.308 [-2.11 to -0.51] | -0.727 [-1.55 to 0.100]
Statistical Analysis 1: Comparison: Placebo vs 1000 mg Epeleuton; Test type: Superiority; p = 0.0763, ANCOVA; LS Mean Difference = -1.308, 95% CI 2-sided [-2.11 to -0.51]
Statistical Analysis 2: Comparison: Placebo vs 2000 mg Epeleuton; Test type: Superiority; p = 0.0058, ANCOVA; LS Mean Difference = -0.727, 95% CI 2-sided [-1.554 to 0.100]

3. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) in Each Treatment Group Leading to Treatment Discontinuation
Description: Subjects with at least 1 TEAE leading to treatment discontinuation
Time Frame: 20 Weeks
Population: The Safety Analysis Set consists of all patients who took at least one administration of study treatment. Patients were analysed according to the treatment actually taken.
Measure: Number; unit: TEAEs
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 31 | 32 | 33
TEAEs | 1 | 0 | 0

4. Secondary Outcome: Change in Serum ALT (Alanine Aminotransferase) From Baseline to Weeks 2, 4, 8 and 12
Description: Change in serum ALT from baseline to weeks 2, 4, 8 and 12.
Time Frame: 12 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 30 | 32 | 31
U/L
  Change from Baseline to Week 2 | -0.4 [-13.3 to 12.4] | -0.1 [-13.0 to 12.8] | -5.8 [-18.2 to 6.6]
  Change from Baseline to Week 4 | -3.4 [-14.9 to 8.2] | 4.0 [-7.6 to 15.7] | -1.9 [-13.0 to 9.3]
  Change from Baseline to Week 8 | -8.7 [-23.1 to 5.7] | -12.7 [-27.1 to 1.6] | -3.8 [-17.4 to 9.9]
  Change from Baseline to Week 12 | -18.3 [-45.3 to 8.8] | -19.2 [-45.3 to 6.9] | -3.8 [-28.7 to 21.0]

5. Secondary Outcome: Change in AST (Aspartate Aminotransferase) From Baseline to Weeks 2, 4, 8, 12 and 16
Description: Change in serum AST from baseline to weeks 2, 4, 8, 12 and 16.
Time Frame: 16 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 30 | 32 | 31
U/L
  Change from Baseline to Week 2 | -5.6 [-22.1 to 10.8] | -4.9 [-21.3 to 11.5] | 4.9 [-11.3 to 21.1]
  Change from Baseline to Week 4 | -4.0 [-12.5 to 4.6] | -1.1 [-9.7 to 7.5] | 2.0 [-6.4 to 10.5]
  Change from Baseline to Week 8 | -4.6 [-13.1 to 3.8] | -9.9 [-18.2 to -1.6] | -0.9 [-9.0 to 7.2]
  Change from Baseline to Week 12 | -13.7 [-28.3 to 0.9] | -11.2 [-25.3 to 2.8] | -3.2 [-17.0 to 10.5]
  Change from Baseline to Week 16 | -8.9 [-35.4 to 17.6] | 7.7 [-18.3 to 33.7] | -4.6 [-32.5 to 23.4]

6. Secondary Outcome: Change in AST:ALT Ratio From Baseline to Weeks 2, 4, 8, 12 and 16
Description: Change in AST: ALT ratio from baseline to weeks 2, 4, 8, 12 and 16.
Time Frame: 16 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 30 | 32 | 31
Ratio
  Change from Baseline to Week 2 | 0.00 [-0.12 to 0.12] | -0.04 [-0.15 to 0.07] | 0.05 [-0.06 to 0.16]
  Change from Baseline to Week 4 | 0.02 [-0.06 to 0.09] | -0.03 [-0.10 to 0.05] | 0.06 [-0.02 to 0.13]
  Change from Baseline to Week 8 | 0.01 [-0.06 to 0.08] | 0.00 [-0.06 to 0.06] | 0.03 [-0.04 to 0.09]
  Change from Baseline to Week 12 | 0.02 [-0.07 to 0.11] | 0.03 [-0.05 to 0.11] | 0.01 [-0.07 to 0.09]
  Change from Baseline to Week 16 | 0.03 [-0.07 to 0.14] | 0.10 [0.01 to 0.19] | 0.02 [-0.08 to 0.13]

7. Secondary Outcome: Change in FIB-4 Index From Baseline to Week 16
Description: Change in FIB-4 Index from baseline to week 16. This index is based on age, platelet count, ALT level, and AST level and will be assessed at Baseline (Visit 2) and week 16 (Visit 10). FIB-4 was calculated using the following formula: FIB4 = (Age (years) x AST (U/L))/(Platelet count (10^9/L) x √ALT (U/L)). A decrease in FIB-4 represents a positive outcome. A FIB-4 Index of <1.45 indicates none to moderate fibrosis and an Index of >3.25 indicates advanced fibrosis.
Time Frame: 16 Weeks
Population: The Full Analysis Set (FAS) includes all randomised patients who received at least one administration of study treatment and have at least one post-baseline measurement for FIB-4 Index.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 24 | 27 | 25
Scores on a scale | -0.109 [-0.398 to 0.181] | 0.114 [-0.196 to 0.424] | -0.068 [-0.384 to 0.248]

8. Secondary Outcome: Change in Non-Alcoholic Fatty Liver Disease (NAFLD) Fibrosis Score (NFS) From Baseline to Week 16
Description: Change in NAFLD fibrosis score (NFS) from baseline to week 16. The NFS is based on age, hyperglycemia, BMI, platelet count, albumin level, and AST/ALT ratio. NFS was calculated using the following formula: NAFLD fibrosis score = -1.675 + 0.037 × age (years) + 0.094 × BMI (kg/m^2) + 1.13 × IFG/diabetes (yes = 1, no = 0) + 0.99 × AST/ALT ratio - 0.013 × platelet (×10^9/l) - 0.66 × albumin (g/dl). A decrease in NFS score represents a positive outcome. An NFS score of <-1.455 indicates no advanced fibrosis and a score of >0.676 indicates liver fibrosis.
Time Frame: 16 Weeks
Population: The Full Analysis Set (FAS) includes all randomised patients who received at least one administration of study treatment and have at least one post-baseline measurement for NFS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 24 | 27 | 25
Scores on a scale | -0.0073 [-0.2653 to 0.2507] | 0.2250 [-0.0529 to 0.5028] | -0.0340 [-0.3149 to 0.2469]

9. Secondary Outcome: Change in ELF (Enhanced Liver Fibrosis Score) From Baseline to Week 16
Description: Change in ELF from baseline to week 16. Enhanced Liver Fibrosis score is an extracellular matrix marker set consisting of tissue inhibitor of metalloproteinases 1 (TIMP-1), amino-terminal propeptide of type III procollagen (PIIINP) and hyaluronic acid (HA). A decrease in ELF score represents a positive outcome. The ELF score was calculated for the instrument based on the following equation: ELF score = 2.494 + 0.846 In (CHA) + 0.735 In (CPIIINP) + 0.391 In (CTIMP-1). An ELF score of less than 7.7 indicates no fibrosis. An ELF score greater than or equal to 9.8 indicates severe fibrosis. An ELF score of 11.3 or greater indicates cirrhosis.
Time Frame: 16 Weeks
Population: The Full Analysis Set (FAS) includes all randomised patients who received at least one administration of study treatment and have at least one post-baseline measurement for ELF.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 25 | 29 | 29
Scores on a scale | 0.24 [-0.09 to 0.56] | 0.10 [-0.19 to 0.39] | 0.01 [-0.29 to 0.31]

10. Secondary Outcome: Change in HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) From Baseline to Weeks 2, 4, 8, 12 and 16
Description: Change in HOMA-IR from baseline to weeks 2,4,8,12,16. Homeostatic model assessment for insulin resistance (HOMA-IR) was assessed as a measure of insulin resistance. HOMA-IR is calculated by multiplying fasting plasma insulin by fasting plasma glucose, then dividing by the constant 405. A decrease in HOMA-IR indicates a positive outcome. HOMA-IR values of greater than 1.9 indicates early insulin resistance and levels above 2.9 indicate significant insulin resistance.
Time Frame: 16 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: HOMA-IR
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 30 | 31 | 31
HOMA-IR
  Change from Baseline to Week 2 | 1.208 [-1.102 to 3.518] | 1.250 [-1.024 to 3.525] | -0.569 [-2.762 to 1.623]
  Change from Baseline to Week 4 | 2.175 [-1.393 to 5.743] | -0.540 [-4.154 to 3.075] | 2.347 [-1.166 to 5.860]
  Change from Baseline to Week 8 | 6.606 [0.563 to 12.649] | 1.817 [-4.280 to 7.913] | 4.283 [-1.707 to 10.273]
  Change from Baseline to Week 12 | -0.045 [-1.769 to 1.680] | 0.00 [-1.677 to 1.678] | -0.258 [-1.858 to 1.343]
  Change from Baseline to Week 16 | -0.393 [-1.310 to 0.524] | -0.326 [-1.234 to 0.582] | -2.037 [-2.912 to -1.162]

11. Secondary Outcome: Change in Adipo-IR (Adipose Tissue Insulin Resistance) From Baseline to Weeks 2, 4, 8, 12 and 16.
Description: Change in Adipo-IR from baseline to weeks 2, 4, 8, 12 and 16. Adipose tissue insulin resistance (Adipo-IR) was assessed as a measure of insulin resistance. Adipo- IR is calculated by multiplying fasting non-esterified fatty acids by fasting insulin. A decrease in Adipo-IR indicates a positive outcome.
Time Frame: 16 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Adipo-IR
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 30 | 31 | 31
Adipo-IR
  Change from Baseline to Week 2 | 9.69 [-6.05 to 25.42] | -5.55 [-21.08 to 9.97] | -10.80 [-25.66 to 4.06]
  Change from Baseline to Week 4 | 24.88 [1.94 to 47.82] | 3.45 [-19.86 to 26.75] | 4.19 [-18.09 to 26.47]
  Change from Baseline to Week 8 | 25.52 [5.86 to 45.18] | 10.40 [-9.28 to 30.07] | 6.63 [-11.79 to 25.05]
  Change from Baseline to Week 12 | 4.20 [-12.46 to 20.86] | -6.28 [-22.88 to 10.32] | -20.66 [-36.35 to -4.97]
  Change from Baseline to Week 16 | 3.66 [-12.54 to 19.86] | -10.68 [-26.80 to 5.43] | -21.07 [-36.44 to -5.69]

12. Secondary Outcome: Change in Hepatic Fat Measured by CAP (Controlled Attenuation Parameter) From Baseline to Week 16.
Description: Change in hepatic fat measured by CAP (controlled attenuation parameter) from baseline to week 16 using FibroScan® 502 Touch model or equivalent. CAP score is measured in decibels per meter (dB/m). A reduction in hepatic fat measured non-invasively by CAP indicates an improvement in hepatic steatosis. CAP scores range from 100 to 400dB/m. 0 to 237 dB/M indicates no hepatic steatosis, 238 to 260 dB/m indicates mild hepatic steatosis, 260 to 290 dB/m indicates moderate steatosis and a CAP score greater than 290 dB/m indicates severe steatosis.
Time Frame: 16 Weeks
Population: The Full Analysis Set (FAS) includes all randomised patients who received at least one administration of study treatment and have at least one post-baseline measurement for hepatic fat measured by CAP.
Measure: Least Squares Mean (95% Confidence Interval); unit: dB/m
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
Number analyzed (Participants) | 27 | 31 | 29
dB/m | -12.3 [-34.4 to 9.9] | -16.3 [-36.8 to 4.1] | -22.4 [-43.0 to -1.8]

ADVERSE EVENTS:
Time Frame: Up to 20 Weeks
Description: An adverse event is any undesirable experience occurring to a patient that has signed the ICF and who has taken their first dose of the study drug, whether or not considered related to the investigational IMP(s). All Adverse Events (AEs) must be recorded in the CRF, defining relationship to IMP and severity. AEs should also be recorded by the Investigator in the patient file/notes.
Arm/Group | Placebo | 1000 mg Epeleuton | 2000 mg Epeleuton
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/32 | 1/33
Other Adverse Events (participants affected / at risk) | 16/31 | 20/32 | 14/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | 1000 mg Epeleuton (N=32) | 2000 mg Epeleuton (N=33)
Pilonidal Cyst (Infections and infestations) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | 1000 mg Epeleuton (N=32) | 2000 mg Epeleuton (N=33)
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 5 | 2
Dizziness (Nervous system disorders) | 0 | 3 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 3
Migraine (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 3 | 0
Blood potassium increased (Investigations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood folate decreased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Faecal volume increased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 1
Fatigue (General disorders) | 1 | 3 | 0
Hyperthermia (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Crystalluria (Renal and urinary disorders) | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 1 | 0 | 0
Endodontic procedure (Surgical and medical procedures) | 0 | 0 | 1
Physiotherapy (Surgical and medical procedures) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT02941549/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT02941549/SAP_001.pdf